CLINICAL TRIAL: NCT06200649
Title: The Effect of Back Massage Applied to Mothers in the Early Postpartum Period on Comfort, Pain, Anxiety, and Physiological Parameters
Brief Title: The Effect of Back Massage Applied to Mothers in the Early Postpartum Period on Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Gamze ŞAHBAZ ÇADIR, Expert Nurse- PhD student, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OUCADIR001
Record Dates: First submitted 2023-01-09; First posted 2024-01-11 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Postpartum Disorder
Keywords: Postpartum Period; Mother; Massage; Comfort; Pain; Anxiety; Physiological Parameters; Nursing
MeSH Terms: conditions — Puerperal Disorders; Pain; Anxiety Disorders | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It will not be clearly stated to the independent statistician which group the intervention and control group participants are in, the groups will be identified with letters as A-B and sent to the statistician for data analysis. The statistical analysis phase of the study will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Massage will be applied to the intervention group by the researcher who has received training in classical massage techniques and has a certificate. The massage will start with effusion (stroking) and will end with effleurage (stroking).
  Baby oil will be used during the massage in order to provide slipperiness and to prevent mothers and babies from being affected by the smell. The oil used will be spread on the back by patting. The massage will last 20 minutes. Post-test data will be obtained by re-filling the forms after 3 hours (6 hours after Normal Birth) for the intervention group to whom massage is applied.
  Interventions: Other: massage
- Control group (No Intervention): No intervention will be made to the control group, and the routine nursing practices of the clinic will continue. Pre-test and post-test will be applied.

INTERVENTIONS:
Other: massage — Massage application; It will be done on the back, which is the five basic massage areas. Massage application will be started with eflorage. The massage will be continued with petrissage by grasping the subcutaneous tissue and muscle layer with the help of thumb and other fingers, starting from the waist circumference. Petrissage will be applied for 5 minutes. After petrissage, the massage was continued with friction movements, which is the other stage. Friction will be applied for 5 minutes. Tapotment will be done after friction. Tapotman will take 5 minutes. After taping, the entire back area will be finished by efflorescence for 2 minutes, just like at the beginning.
  Arms: Intervention Group

SUMMARY:
In the literature, there are separate studies on massage, comfort, anxiety, and physiological parameters for massage practice, but there are no studies that measure the physiological parameters of comfort, pain, anxiety, blood pressure, pulse, fever, oxygen saturation, respiratory rate in the early postpartum period. In this study, the effect of back massage applied to mothers in the early postpartum period on comfort, pain, anxiety and physiological parameters will be examined.

If it is determined that the massage application, which is easy to apply and effective, has a positive effect on physiological parameters such as comfort, pain, anxiety and blood pressure, pulse, fever, oxygen saturation, respiratory rate, as well as other parameters measured in the postpartum period, it can be used in the field of application.

This is where the originality of our work comes from. For this reason, it is aimed to contribute to the literature with this study.

DETAILED DESCRIPTION:
For this purpose, pharmacological and non-pharmacological interventions should be made for these conditions seen in the postpartum period. It is possible to increase the quality of health care, to make a difference in patient care results and clinical practices, to increase patient satisfaction rates and to standardize care, especially by using non-pharmacological methods whose effectiveness has been proven by health professionals. As a matter of fact, studies indicate that postpartum women who receive effective nursing care are highly satisfied (88-90%) with the care services they receive. It is important for health professionals to follow current and high-evidence studies, conduct research on their own development and participate in in-service programs in order to increase the quality of health care. There are many practices such as aromatherapy and yoga applied in the postpartum period. Massage is one of them.

Massage is a process applied systematically to the soft tissues of the body, providing relaxation and mental relief. Theoretically, massage stimulates peripheral receptors in the skin. The stimuli reach the brain via the spinal cord and provide general relaxation. Massage reduces cortisol, adrenaline and noradrenaline levels by regulating the autonomic nervous system. The amygdala may also modulate neural activity in the forebrain and control network. The pressure in massage application increases blood circulation and lymphatic drainage, causing changes in heart rate and blood pressure. This non-pharmacological method helps to increase comfort by relaxing the muscles, increase the release of endorphins, urinary serotonin and dopamine, decrease salivary and urinary cortisol levels, reduce pain and edema, and treat psychological disorders such as depression and anxiety. If it is determined that the massage application, which is easy to apply and effective, has a positive effect on physiological parameters such as comfort, pain, anxiety and blood pressure, pulse, fever, oxygen saturation and respiratory rate, as well as other parameters measured in the postpartum period, it can be used in the application area. This is where the originality of our work comes from. For this reason, it is aimed to contribute to the literature with this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over
* Vaginal delivery
* In the first 24 hours after birth
* First born
* Having no difficulty in sitting
* Written / verbal communication can be established
* At least primary school graduate
* Not having any problems during mother's pregnancy
* Not diagnosed with any psychiatric disease
* Wound, infection, mass etc. on the back. non
* Vascular and cardio-thoracic diseases, non-skin diseases
* Women who agree to participate in the study will be taken into the sample

Exclusion Criteria:

* Being under 18 years old
* Giving birth by cesarean section
* Receiving controlled analgesia after normal delivery
* Women with a psychiatric diagnosis will not be included in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-06-09 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Postpartum Comfort Scale | two year
  Postpartum Comfort Scale consists of 34 items and is a 5-point Likert type. For each item, wording and scoring ranging from "completely agree" (5 points) to "strongly disagree" (1 point) were used. Accordingly, the lowest score from the scale can be 34 and the highest score can be 170. Positive expressions in the scale (1, 2, 3, 5, 7, 11, 14, 15, 18, 19, 20, 23, 24, 25, 31, 32) are coded as 1: I strongly disagree - 5: I completely agree. In the negative items (4, 6, 8, 9, 10, 12,13, 16, 17, 21, 22, 26, 27, 28, 29, 30, 33, 34), it is reversed as "I totally disagree, 5 I totally agree, 1". coded. The average value is determined by dividing the total score obtained from the scale by the number of items and the result is shown in the 1-5 distribution. Basically, low comfort is expressed as 1 and high comfort is expressed as 5.

SECONDARY OUTCOMES:
Visual Analogue Scale | two year
  The Visual Analog Scale is a one-dimensional scale frequently used to determine people's pain levels. The patient makes a mark on a horizontal or vertical ruler of 10 cm or 100 mm, depending on where he sees fit according to the severity of pain. In the result evaluation, 0 cm was stated as "no pain", 0.5 cm-3 cm was stated as "mild pain", 3.5 cm-6.5 cm was stated as "moderate pain", and 7-10 cm was stated as "severe pain". As the score increases, the pain level increases.

OTHER OUTCOMES:
Physiological Parameters Form | two year
  Physiological parameters are important indicators in the management of the postpartum period and in determining the treatment protocol. Blood pressure, body temperature, heart rate, respiratory rate and oxygen saturation, which are stated as basic life parameters, are parameters that indicate the health status of the person. For this purpose, the Physiological Parameters Form includes blood pressure, body temperature, heart rate, oxygen saturation and respiratory rate.
determining postpartum anxiety | two year
  The scale is a four-point Likert type and consists of two parts: State-Trait Anxiety Inventory and Trait Anxiety Inventory. There are 20 questions in each section. For the State Anxiety Scale, "Not at all" is 1, "Somewhat" is 2, "A lot" is 3, "Completely" is 4; For the trait anxiety inventory, "Almost never" is marked as 1, "Sometimes" is marked as 2, "Most of the time" is marked as 3, and "Almost always" is marked as 4. Scales range from 20 to 80. High scores indicate high anxiety. The scale includes reverse and true expressions. When scoring reverse expressions, those with a weight of 1 are given a score of 4; Those with a weight value of 4 are converted to 1.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Şahbaz Çadır, PHD STUDENT, Principal Investigator — Ordu University; Nülüfer Erbil, Prof. Dr., Study Director — Ordu University
Locations (1):
- Kahramanmaraş, Necip Fazıl City Hospital Gynecology and Pediatrics Additional Service Building, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No